CLINICAL TRIAL: NCT00459927
Title: Prospective, Controlled Clinical Trial of a Novel Hemostatic Sealant Versus Electrocautery Hemostasis and Coblation Dissection in Patients Undergoing Tonsillectomy
Brief Title: Comparison of Floseal Hemostasis Tonsillectomy With Coblation Tonsillectomy and Cautery Hemostasis Tonsillectomy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Siri Sunderi Cheng, MD, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CN-06JGott-01-B
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Adenotonsillar Hypertrophy; Tonsillitis; Obstructive Sleep Apnea
Keywords: Adenotonsillectomy; Coblation tonsillectomy; Floseal
MeSH Terms: conditions — Tonsillitis; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Floseal tonsillectomy
Device: Coblation tonsillectomy

SUMMARY:
The purpose of this study is to evaluate a new method of hemostasis, floseal gel, in tonsillectomy and adenoidectomy, with the goal of decreasing post operative and intraoperative morbidity.

DETAILED DESCRIPTION:
Blood loss and postoperative morbidity following adenotonsillectomy in children can be significant. The current technique for performing a tonsillectomy is "cold steel tonsillectomy" with electocautery hemostasis and a newer technique of coblation tonsillectomy. Postoperative pain has been shown to be increased in patients undergoing extensive electrocautery, with less pain seen in patients undergoing coblation tonsillectomy. The purpose of the study is to evaluate the clinical efficacy and complications of Floseal matrix hemostatic sealant for use in patients undergoing adenotonsillectomy compared with two other currently used techniques.

The study is a prospective, controlled clinical trial comparing Floseal hemostasis in "cold steel" knife dissection tonsillectomy with cautery hemostasis in "cold steel" knife dissection tonsillectomy and coblation tonsillectomy in a pediatric population. All children under the age of 18 without previous documented coagulopathy scheduled to undergo tonsillectomy will be offered enrollment in the study. Informed consent will be obtained from the patient's legal guardian. The goal of this study is to determine if Floseal reduces intraoperative blood loss, time to hemostasis, and postoperative morbidity in patients undergoing tonsillectomy compared with two other commonly used methods. Also, we wish to evaluate the complication rates following Floseal administration compared to those of electrocautery and coblation.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years old scheduled for a routine adenotonsillectomy

Exclusion Criteria:

* Down syndrome
* Craniofacial abnormality

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-07

PRIMARY OUTCOMES:
Intraoperative: Procedure time, hemostasis time, difficulty of hemostasis, blood loss | intraoperative period
Postoperative: Amount of pain medication required (day 1-14), subjective pain score, postoperative day # for returning to a normal diet and normal activity | postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Gottschall, M.D., Principal Investigator — Kaiser Permanente